CLINICAL TRIAL: NCT04709991
Title: Comparison of Lower Limb Endovascular Interventions With and Without the EndoNaut Workstation
Acronym: COMPAR-MI
Status: Completed | Type: Observational
Sponsor: Therenva (Industry)
Collaborators: CH Libourne (Unknown)
Responsible Party: Sponsor
Other Study IDs: 001
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Endovascular Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Procedures with EndoNaut
  Interventions: Procedure: Endovascular procedure
- Procedures without Endonaut
  Interventions: Procedure: Endovascular procedure

INTERVENTIONS:
Procedure: Endovascular procedure — Creation of a bone and arterial panorama using EndoNaut® software. The routine care procedure begins with staged injections of contrast medium to provide a map of the lesions. The lesions are then treated by angioplasty with or without stenting.

SUMMARY:
To demonstrate that the use of EndoNaut for endovascular procedures on the femoropopliteal axis has a clinical impact for the patient (decrease in irradiation and the volume of contrast product) as well as for nursing staff (reduction in irradiation) compared to procedures performed without EndoNaut.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) is characterized by a narrowing of the size of arteries, which resulting in a loss of hemodynamic load. Endovascular (or percutaneous) procedures performed at the infrainguinal level (axefemoro-popliteal) are very common in affected patients. Therenva offers a complete and consistent lightweight navigation solution (EndoNaut®) based on artificial intelligence (AI) algorithms, and providing technology accessible to all operating rooms for PAD procedures. The aim of this study is to demonstrate that the use of EndoNaut for endovascular procedures on the femoropopliteal axis has a clinical impact for the patient (decrease in irradiation and the volume of contrast product) as well as for nursing staff (reduction in irradiation) compared to the procedures performed by EndoNaut.

ELIGIBILITY:
Inclusion Criteria:

* Patients with peripheral arterial disease of the lower limbs, all clinical stages, lesions of the femoro-popliteal stage and candidates for endovascular treatment of these lesions.
* Major patients
* Patients not opposed to their participation in the study

Exclusion Criteria:

- Patients requiring conventional surgical revascularization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic occlusive arthritis of the Lower Limbs with lesions on the femoro-popliteal stage and candidates for endovascular treatment of these lesions.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Volume of contrast product used during the routine care procedure (ml) | 1 day At enrollment
  Volume are reported in mL
Irradiation parameters: evaluation of the Fluoroscopy duration (min) | 1 day At enrollment
  Parameter given by the X-ray imaging device
Irradiation parameters: dose-area quantification (mGy/m2) | 1 day At enrollment
  Parameter given by the X-ray imaging device
Irradiation parameters: measurement of air Kerma (mGy) | 1 day At enrollment
  Parameter given by the X-ray imaging device

CONTACTS AND LOCATIONS:
Locations (1):
- CH Libourne, Libourne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Caradu C, Stenson K, Houmaida H, Le Ny J, Lalys F, Ducasse E, Gheysens B. EndoNaut two-dimensional fusion imaging with a mobile C-arm for endovascular treatment of occlusive peripheral arterial disease. J Vasc Surg. 2022 Feb;75(2):651-659.e1. doi: 10.1016/j.jvs.2021.08.069. Epub 2021 Sep 10. PMID 34509588